CLINICAL TRIAL: NCT04896905
Title: Rehabilitation After Covid19-Clinical Results and Predictive Factors for Rehabilitation Outcomes
Brief Title: Rehabilitation After Covid19-Clinical Results and Predictive Factors
Status: Completed | Type: Observational
Sponsor: Klinik Valens (Other)
Responsible Party: Principal Investigator, Stefan Bachmann, Chief Medical Officer, Clinical Professor, Klinik Valens
Other Study IDs: Covid19_2020
Record Dates: First submitted 2021-05-19; First posted 2021-05-21 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: Covid19
Keywords: Covid19; Sars-CoV-2; Rehabilitation; Outcome; Predictive factors
MeSH Terms: conditions — COVID-19 | interventions — Rehabilitation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Isolation group with active Covid19: Patients assigned to rehab which had to be treated in isolation wards dur to active disease
  Interventions: Other: Rehabilitation
- Post-Covid-group: Patients assigned to rehab after active disease, still having restrictions in activity and particiaption
  Interventions: Other: Rehabilitation
- Control group: Pateints assigned to rehabilitation in the same time period without any signs of Sars-coV-2 infection
  Interventions: Other: Rehabilitation

INTERVENTIONS:
Other: Rehabilitation — Rehabilitative procedures in isolation ward

SUMMARY:
The aim of the study is to gain insight into the rehabilitation process and predictive factors for the outcome after rehabilitation in three patient groups:

1. SARS-CoV-2-positive patients in the isolation ward
2. Post-Covid-19 patients
3. Control group; matched for gender, age and co-morbidity

ELIGIBILITY:
Inclusion Criteria:

* Patients assigned to rehab
* Written informed consent

Exclusion Criteria:

* not able to fill in questionnaires in German

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients referred to rehabilitation between March and June 2020 either with active Covid19, post-Covid-State oor other indications for inpatient rehab (eg. muskuloskelettal, cancer, pulmonary diseases not related to Covid19)
Sampling Method: Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-05-18 (Actual)

PRIMARY OUTCOMES:
Mobility | Measurements done at entry and at discharge of rehabilitation (time between: 4- 6 weeks)
  Timed Up and Go-Test TUG (Seconds; less=better, normal <10 Sec.)
Functional Independence Measurement-Level (FIM) | Measurements done at entry and at discharge of rehabilitation (time between: 4- 6 weeks)
  FIM at entry and discharge (min 18, max 126 points; higher level= better functioning; )
Promis-10 (Promis= Patient reported outcome measurement information system) | Measurements done at entry and at discharge of rehabilitation (time between: 4- 6 weeks)
  Level of patient self rated functioning in daily activities (higher level= better self related functioning)
Quality of life | Measurements done at entry and at discharge of rehabilitation (time between: 4- 6 weeks)
  EQ5D- VAS (0-100; higher level = better quality of life)

CONTACTS AND LOCATIONS:
Overall Officials: Steffi Petzold, MMed, Principal Investigator — Kliniken Valens; Roisin Carney, PT, cand MSc, Principal Investigator — Kliniken Valens
Locations (1):
- Rehabilitationszentrum Klinik Valens, Valens, Canton of St. Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: No